CLINICAL TRIAL: NCT04107025
Title: Effects of a Legal Support Program on Women Experiencing Domestic Violence: Help Intervention Study
Brief Title: Effects of a Legal Support Program on Women Experiencing Domestic Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NMP/07845
Record Dates: First submitted 2019-09-24; First posted 2019-09-27 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-09

CONDITIONS: Domestic Violence; Anxiety; Depression; Stress
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): As part of the intervention, along with legal opinions, advise and support, participants were provided counselling support during their time to help survivors with trauma of legal proceedings.
  Interventions: Other: HELP
- Usual Care (No Intervention): Participants were scheduled for legal consultancy only.

INTERVENTIONS:
Other: HELP — Individual counseling were given to each intervention group participant. They were assisted with safety, emotional and mental support and referrals for health and financial assistance. Participants were also given handout to manage anxiety and panic situations during the legal procedures.
  Arms: Intervention

SUMMARY:
Intimate partner violence (IPV) is a major public health concern. Worldwide, 1 in 3 women have experienced domestic abuse/ violence in their lifetime. In most cases, family lawyers, advocates are first contact before the police. If the children are involved, finding the legal options become the priority for women before leaving the abuser.

The purpose of this study was to compare the effectiveness of the HELP (Health, Education Legal Support Program) intervention among IPV survivors.

ELIGIBILITY:
Inclusion Criteria:

* Female survivors of Intimate Partner Violence
* 18 years old or older
* Gives informed consent

Exclusion Criteria:

* Diagnosed mental health condition
* Terminally ill
* Chronic condition
* On psychiatric medication
* Sexual assault

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female survivors of domestic violence
Enrollment: 56 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-12 (Actual)

PRIMARY OUTCOMES:
Anxiety | Change from baseline anxiety symptoms at 4 weeks
  Anxiety symptoms were assessed using the Hospital Anxiety Depression Scale
Depression | Change from baseline depression symptoms at 4 weeks
  Depression symptoms were assessed using the Hospital Anxiety Depression Scale
Stress | Change from baseline stress symptoms at 4 weeks
  Perceived Stress Scale was used to assess stress symptoms

SECONDARY OUTCOMES:
Self esteem | Change from baseline self esteem at 4 weeks
  Rosenberg's Self-Esteem Scale was used to measure self esteem

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Warwick Research Services; Anurag Sharma, MPhil, Study Chair — Patan Girls College; Rekha Khandelwal, PhD, Principal Investigator — NMP Medical Research Institute, India
Locations (2):
- India (2):
  - Gyansanjeevani, Būndi, Rajasthan
  - Gyansanjeevani, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided